CLINICAL TRIAL: NCT00199966
Title: A Pilot Study Of Safety And Effectiveness For Depakote ER In Pediatric Bipolar Disorder
Brief Title: Safety And Efficacy Study Of Depakote ER To Treat Pediatric Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHW 03/163, HRRC 539-03
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Pediatric Bipolar Disorder; Depakote ER
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Divalproex sodium extended release

SUMMARY:
The purpose of this research is to compare how safely and how well this medicine works in treating children and teenagers between the ages of 6 and 17 years with a diagnosis of Bipolar Disorder.

DETAILED DESCRIPTION:
There is no accepted, well-studied treatment for Pediatric Bipolar Disorder and treatment has often followed from adult studies. The primary objectives for this study are to determine if subjects can safely and easily be switched from divalproex sodium to Depakote ER and to determine if Depakote ER is both safe and effective for pediatric patients with Bipolar I or II. Secondary objectives include determining the serum levels of valproic acid 20 hours after administration of Depakote ER at a steady rate and determining if co-administration of stimulants will effect the serum levels of valproic acid. Thirty subjects, ages 6-17 years, with a diagnosis of Bipolar I or II who are currently asymptomatic, according to a score of less than 10 on the Young Mania Rating Scale, or who desire to change to once daily dosing, or desire to change because of the likelihood of decreased side-effects, will be recruited from our clinic and the community. If subjects have completed baseline evaluations (including diagnostic confirmation), labs, and rating scales and are still eligible to participate, subjects will be switched in one night from twice-a-day divalproex sodium (DVP) to divalproex sodium extended release (DVP ER).

The potential benefits of the research are that new information will be added to the field of child and adolescent psychiatry and the possibility that the medication change may result in improved symptoms of mania or side effects of medications related to peak and trough levels. The potential benefits of this study outweigh the possible risks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bipolar I or II confirmed by K-SADS and clinical interview.
* Ages 6 to 17 years 11 months.
* YMRS score of <10, this is consistent with minimal symptoms of mania. Or a desire to change medications due to a simplified dosing schedule or to reduce unwanted side effects of divalproex sodium.
* Ability and willingness of subject and parent(s)/guardian(s) to provide informed written assent/consent.

Exclusion Criteria:

* Diagnosis of: Pervasive Developmental Disorders, Schizophrenia spectrum disorders, Obsessive Compulsive Disorder.
* Concurrent medical conditions requiring medication or that are unstable.
* Current suicidal thoughts.
* Recent suicidal behavior.
* Pregnancy or sexually active female not using a reliable form of contraception.
* Previous inadequate response to DVP ER.
* Known hypersensitivity to DVP or DVP ER.
* Recent inpatient hospitalization for suicidality or homicidality, (last 6 months).
* Subjects who are clinically stable and not suffering significant side effects on their current medical regimen.
* Use of antidepressants within the last 2 weeks, 4 weeks for fluoxetine.
* Recent (last 3 months) substance abuse or dependence. Urine drug screen will be obtained if a question arises.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30
Dates: Start 2003-12; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Young Mania Rating Scale (YMRS), rate at baseline, Week 2,4,6,&8

SECONDARY OUTCOMES:
Kiddie version of the Schedule for Affective Disorders and Schizophrenia (KSADS), assessed at baseline only.
Child Depression Rating Scale (CDRS), rate at baseline through Week 8.
Clinical Global Impression: Improvement and Severity (CGI), for mania, depression and ADHD. Rate from baseline through Week 8.
Conner's Parent and Teacher Rating Scales (CRS). Rate from baseline through Week 8.
Side Effect For Children & Adolescents (SEFCA). Rate from baseline through Week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Russell E Scheffer, MD, Principal Investigator — Medical College of Wisconsin; Children's Hospital of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States